CLINICAL TRIAL: NCT07397975
Title: A Prospective Multicenter Study for Relapse Risk Assessment Through Language Analysis in Individuals With Psychosis
Brief Title: Speech-based Assessment of Relapse Risk in People With Psychosis
Acronym: TRUSTING-WP4
Status: Recruiting | Type: Observational
Sponsor: Philipp Homan (Other)
Responsible Party: Sponsor-Investigator, Philipp Homan, Prof. Dr. med. univ. Philipp Homan, PhD, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: TRUSTING-WP4-Obs_EK2025-01177
Record Dates: First submitted 2026-01-22; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Psychotic Disorder
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- At risk of relapse: Individuals at risk of psychotic relapse
  Interventions: Other: Weekly online speech assessments via a smartphone app collect speech and self-report data. Recordings are securely transferred and analyzed by an AI-based backend to calculate relapse risk scores.
- Healthy controls: Healthy participants will be used as controls
  Interventions: Other: Weekly online speech assessments via a smartphone app collect speech and self-report data. Recordings are securely transferred and analyzed by an AI-based backend to calculate relapse risk scores.

INTERVENTIONS:
Other: Weekly online speech assessments via a smartphone app collect speech and self-report data. Recordings are securely transferred and analyzed by an AI-based backend to calculate relapse risk scores. — The intervention is a weekly online assessment of speech, to detect subtle characteristics of psychotic speech. These recordings are made through a speech data collection tool: a smartphone app with implemented tasks for the collection of behavioral response data (speech and self-report). Data is then transferred to a safe repository (TSD) to be analysed by an AI-based speech data analysis algorithm: a backend system will run the predictor code to calculate automatic relapse risk scores.

SUMMARY:
This observational, multinational study assesses the feasibility of speech and self-report data collection across six languages for Artificial Intelligence (AI)-driven relapse risk estimation in psychosis. Over 12 months, patients at risk of relapse and healthy controls will provide weekly speech recordings and self-report data for automated analysis. Risk scores will be stored but not shared with treating clinicians. Independent clinical evaluations ensure data quality and validation. The study lays the foundation for future Clinical Decision Support System (CDSS) research and explores novel speech markers for relapse prediction while minimizing participant burden.

DETAILED DESCRIPTION:
This project follows a prospective, exploratory, observational design with a non-randomized, two-arm structure, including a group of individuals with psychosis at risk of relapse and a healthy control group. As a multicenter, international research project, it will assess the usability and feasibility of speech data collection across 6 different languages (English, German, French, Dutch, Czech and Turkish) and healthcare systems, ensuring its applicability in diverse clinical environments.

Speech and self-report data will be collected weekly for a year using a finalized smartphone application, ensuring consistency and feasibility in real-world clinical settings. The recordings will be securely transferred to an external platform for AI-based analysis, preventing any direct impact on clinical decision-making and maintaining the study's observational nature.

To ensure data integrity and reliability, a Human-in-the-Loop (HITL) quality control process is implemented after each speech recording session:

Initial Data Review: a designated reviewer (HITL1) checks the audio quality and accuracy of automated transcripts stored securely in the Trusted Secure Database (TSD) system in Norway. They correct transcription errors and flag anomalies such as poor audio quality to maintain data accuracy for analysis.

Risk Assessment and Decision Suggestion: a second reviewer (HITL2) evaluates the data by: (i) assessing speech characteristics relevant to relapse risk based on raw response data and performance scores (e.g., story recall accuracy); (ii) providing an independent relapse risk estimate, without access to the automated AI-generated risk assessment, (iii) classify the participant as belonging to either the psychosis or healthy control group, and (iv) suggesting a clinical decision, which is recorded for research purposes but not shared with the treating clinician.

Apart from this Fast Diagnostic Loop, where a clinical decision will be made, an exploratory component will be incorporated to identify and validate new speech markers associated with relapse. This New Marker Discovery Loop will involve the search of additional speech features associated with relapse beyond the standard markers. The goal is to discover novel speech markers that may improve our understanding of relapse mechanisms and potentially serve as predictive or diagnostic tools for future clinical use.

For the 1-year follow-up period, participants will attend a total of three study visits. These visits will occur at the following time points: Visit 0: Baseline visit, Visit 1: 6 months post-baseline (±10 days), and Visit 2: 12 months post-baseline (±10 days). During these visits, participants from both groups will undergo assessments aiming to evaluate the usability and trustworthiness of the procedure and to assess various functional and quality-of-life outcomes.

ELIGIBILITY:
Healthy participants Inclusion Criteria:

* Between 18 and 65 years old.
* Subjects must be able to provide informed consent (IC).
* Participants must have provided signed informed consent prior to enrollment.
* Participants should not take prescription drugs regularly.
* Native or equivalent fluency in speaking and understanding one of the following languages: English, German, Dutch, French, Czech or Turkish.
* Ability to have access to a smartphone and be capable of using a mobile app for speech-based data collection.
* Must be able to comply with the study schedule and procedures.

Healthy participants Exclusion Criteria:

* Any history of major diseases (e.g., cardiovascular, neurological, metabolic, renal, hepatic, respiratory or speech disorders).
* Recreational drug use or psychiatric disorders due to use of alcohol.
* Depression, anxiety, or other psychiatric disorders.
* Family history of depression, anxiety, or other psychiatric disorders.
* Individuals who are not able or willing to understand the purpose and details of the study.

Individuals with psychosis Inclusion Criteria:

* Between 18 and 65 years old.
* Diagnoses include psychotic disorders (schizophrenia, schizoaffective disorder, schizophreniform disorder, acute psychosis, bipolar disorder with psychotic symptoms, psychosis not otherwise specified).
* First visit must be during remission phase (baseline measurement).
* Current positive symptoms rated 3 (mild) or lower on all of these Brief Psychiatric Symptom Scale (BPRS) items: hallucinatory behavior, unusual thought content, conceptual disorganization.
* Must be able to comply with the study schedule and procedures.
* Subjects must be able to provide IC.
* Participants must have provided signed informed consent prior to enrollment.
* Native or equivalent fluency in speaking and understanding one of the following languages: English, German, Dutch, French, Czech or Turkish.
* Ability to have access to a smartphone and be capable of using a mobile app for speech-based data collection.

Individuals with psychosis Exclusion Criteria:

* Severe comorbid speech disorders (aphasia or severe stuttering) that prevent adequate speech recording.
* Individuals who are not able or willing to understand the purpose and details of the investigation.

Citizens with psychiatric or somatic comorbidity, drug- or alcohol abuse will be allowed to participate, so that the sample will reflect the general population of citizens with psychosis and the study's endpoints will be generalizable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants at risk of relapse will be recruited from clinical settings while in a stable phase of partial or full remission. Depending on the site, eligible individuals may be either inpatients nearing discharge or outpatients under ongoing care. If the treating clinician considers the patient's mental state sufficiently stable, the study information and consent process may be initiated during inpatient care, prior to discharge. For outpatients, participants may be contacted by phone, or the study can be presented during routine outpatient or day clinic visits.
  Healthy participants will be recruited through community outreach, advertisements, and volunteer registries from universities and hospitals. healthy participants will be selected to match individuals with psychosis based on key characteristics such as age and sex in each site.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: User adherence | From enrollment to the end of the study at 12 months
  Proportion of users adhering to their allocated tasks. Task completion is automatically assessed for each user. A user is regarded as adherent, if they complete at least 33% of their tasks across all sessions.
Feasibility: Transcription quality | From enrollment to the end of the study at 12 months
  Proportion of users for which high quality transcripts are produced. Transcription quality is measured by the Word Error Rate (WER) between Automated Speech Recognition (ASR) and human corrected transcripts. A user with an overall WER of at most 35% is regarded as having high quality transcripts
Feasibility: Usability of recordings | From enrollment to the end of the study at 12 months
  Proportion of recordings that can be used by the AI algorithm. Usability of each record is assessed by HITL reviewers based on the three questions (i) has the user interpreted the question correctly, and (ii) is the audio (at least partially) audible and (iii) comprehensible. The three questions must both be answered with yes for the recording to be usable
Overall system usability | 6 months and 12 months
  Proportion of users rating the app as usable. Usability is evaluated using the System Usability Scale (SUS), providing a standardized usability score (range 0-100) based on a 10-item questionnaire. We regard a score of at least 70 as usable.
Performance of the monitoring system for relapse prediction | From enrollment to the end of the study at 12 months
  Assessed by the Area Under the Receiver Operating Characteristic Curve (AUC). Thresholds for relapse prediction will be explored as part of the analysis

SECONDARY OUTCOMES:
Provider-perceived usability and usefulness | 6 months and 12 months
  Provider-perceived usability and usefulness of the app will be assessed using the mHealth App Usability Questionnaire (MAUQ - Provider version). Scores will be reported by domain and overall
Relapse Outcome 1 | 6 months and 12 months
  Relapse rate, defined as the proportion of participants experiencing at least one relapse (rehospitalization) during the study period.
Relapse Outcome 2 | From enrollment to the end of the study at 12 months
  Human-in-the-loop (HITL) relapse risk estimates and relapse incidence: HITL risk scores (range 0-1) will be categorized into low (0-0.2), medium (>0.2-0.6), and high (>0.6) risk levels. Descriptive analyses will assess the proportion of relapses within each category.
Relapse Outcome 3 | From enrollment to the end of the study at 12 months
  Clinical decision support system (CDSS) relapse risk estimates and relapse incidence: CDSS risk scores (range 0-1) will be categorized into low, medium, and high risk using the same thresholds. Descriptive analyses will assess relapse proportions per category.
Relapse Outcome 4 | From enrollment to the end of the study at 12 months
  Predictive performance of HITL relapse risk estimates will be evaluated using the area under the curve (AUC), with exploratory assessment of prediction thresholds.
Relapse Outcome 5 | From enrollment to the end of the study at 12 months
  Concordance between CDSS and HITL relapse risk estimates will be assessed by evaluating the level of agreement between algorithm-based and clinician-based risk scores.
Recordings Outcome 1 | From enrollment to the end of the study at 12 months
  Number of recordings per participant across all sessions.
Recordings Outcome 2 | From enrollment to the end of the study at 12 months
  Interpretation of question: has the user interpreted the question correctly? Yes or no. Per recording.
Recordings Outcome 3 | From enrollment to the end of the study at 12 months
  Audibility of audio: is the audio (at least partially) audible? Yes or no. Per recording.
Recordings Outcome 4 | From enrollment to the end of the study at 12 months
  Comprehensibility of audio: is the audio (at least partially) comprehensible? Yes or no. Per recording
Speech-based features | From enrollment to the end of study at 12 months.
  Exploratory comparison analysis of speech-based features extracted using tools such as Prosogram or openSMILE.
Text-based features Outcome 1 | From enrollment to the end of the study at 12 months.
  In addition, robust text-based features like speech rate and pause rate will be derived using common Python libraries for Natural Language Processing (NLP) like NLTK and spaCy.
Text-based features Outcome 2 | From enrollment to the end of the study at 12 months
  WordNet will be used to analyze correctness of responses where appropriate (fluency task, story recall task, adapted Stroop task).
Neuroimaging-based features Outcome 1 | 6 months and 12 months
  Exploratory comparison analysis of features extracted from structural magnetic resonance imaging (sMRI) data.
Neuroimaging-based features Outcome 2 | 6 months and 12 months
  Exploratory comparison analysis of features extracted from functional magnetic resonance imaging (fMRI) data.
Neuroimaging-based features Outcome 3 | 6 months and 12 months
  Exploratory comparison analysis of features extracted from Diffusion Tensor Imaging (DTI) data.
Social and occupational function of participants Outcome 1 | Baseline, 6 months and 12 months
  Quality of life assessed with Quality of Life Scale (QoL). Assessed only in participants at risk of relapse
Social and occupational function of participants Outcome 2 | 6 months and 12 months
  Global Assessment of Functioning Scale (GAF): measures how much a person's symptoms affect their day-to-day life on a scale of 0 to 100. Assessed only in participants at risk of relapse
Social and occupational function of participants Outcome 3 | 6 months and 12 months
  Social and Occupational Functioning Assessment Scale (SOFAS): a global rating of current social and occupational functioning with scores ranging from 0 to 100. It differs from GAF by focusing on social and occupational functioning independent of the overall severity of the individual's psychological symptoms. Assessed only in participants at risk of relapse
Social and occupational function of participants Outcome 4 | 6 months and 12 months
  Number of psychiatric admissions. Assessed only in participants at risk of relapse
Social and occupational function of participants Outcome 5 | 6 months and 12 months
  Duration (in weeks) of psychiatric admissions. Assessed only in participants at risk of relapse
Social and occupational function of participants Outcome 6 | 6 months and 12 months
  Rates of self-harm (including suicide, suicide attempts and aggressive incidents) assessed with the Social Dysfunction & Aggression Scale (SDAS). Assessed only in participants at risk of relapse
Social and occupational function of participants Outcome 7 | 6 months and 12 months
  Positive and Negative Syndrome Scale (PANSS): measure the prevalence of positive and negative syndromes in schizophrenia. Scores will be reported by dimension (positive, negative, and general psychopathology) and overall. Assessed only in participants at risk of relapse

CONTACTS AND LOCATIONS:
Locations (7):
- National Institute of Mental Health, Klecany, Czechia
- Newcastle Hospital and RCSI University of Medicine and Health Sciences, Greystones, Wicklow, Ireland
- University Medical Center Groningen, Groningen, Netherlands
- The Arctic University of Norway, Tromsø, Norway
- Switzerland (2):
  - University Hospital Geneva and University of Geneva, Geneva, Chêne-Bourg
  - Psychiatric University Hospital Zurich and University of Zurich, Zurich
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No